CLINICAL TRIAL: NCT06417021
Title: The Position of the Ultrasound Machine in the Placement of the Central Venous Catheter: a Randomized Controlled Study
Brief Title: Ergonomics in Ultrasound Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 25148/2024
Record Dates: First submitted 2024-04-09; First posted 2024-05-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Procedural Complication; Competence
Keywords: Central Venous Access; Ultrasound; Ergonomics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A clip of the ultrasound procedure will be saved and reviewed by a blind assessor that will value the quality of the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frontal position of Ultrasound machine (Ergonomic group) (Other): Participants will simulate a CVC positioning keeping the ultrasound machine facing them
  Interventions: Other: Frontal Ultrasound Machine
- Lateral position (90°) of Ultrasound machine (No Ergonomic group) (Other): Participants will simulate a CVC positioning keeping the ultrasound machine in a lateral position on the same side of the needle.
  Interventions: Other: Lateral Ultrasound Machine

INTERVENTIONS:
Other: Frontal Ultrasound Machine — Ultrasound machine will be placed in a frontal position
  Arms: Frontal position of Ultrasound machine (Ergonomic group)
Other: Lateral Ultrasound Machine — Ultrasound machine will be placed in a lateral position
  Arms: Lateral position (90°) of Ultrasound machine (No Ergonomic group)

SUMMARY:
The study will compare two different positions of the ultrasound machine during simulated CVC positioning.

The position of the ultrasound machine will be randomized. Group A will perform the procedure with the ultrasound monitor facing them, while subjects randomized to group B will perform the procedure with the ultrasound machine positioned at a 90° angle to their visual axis.

DETAILED DESCRIPTION:
We will recruit medical trainees affiliated with the 'Anesthesia and Intensive Care' and 'Emergency Medicine' schools. Data collected for each participant will include: age, gender, specialty school, year of specialization training, expertise in using ultrasound for ultrasound-guided procedures. Once informed consent is obtained, subjects will be divided through simple randomization (a list generated in advance with Excel and subjected to the opaque envelope method) into two groups: A and B. All subjects will be asked to perform CVC placement using the simulator through an 'oblique in-plane' approach. Subjects randomized to group A will perform the procedure with the ultrasound monitor facing them, while subjects randomized to group B will perform the procedure with the ultrasound machine positioned at a 90° angle to their visual axis.

ELIGIBILITY:
Inclusion Criteria:

* 'Anesthesia and Intensive Care' and 'Emergency Medicine' residents
* Informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Time to correct CVC position | baseline
  Investigators will measure time needed to correctly perform the procedure in seconds. The chronometer will be started when the participant takes the ultrasound probe and will be stopped when the guidewire will be correctly placed

SECONDARY OUTCOMES:
Needle tip visualization | baseline
  Procedure will be recorded as a clip in ultrasound machine. A blind assessor will evaluate the clip using the following scale (1-During the advancement of the needles, only the distortion of the tissue could be observed.
  2-Only the tip of the needle was visible. 3-The tip of the needle was visible throughout the advancement, but the body of the needle was only partially visible.
  4-The needle was completely visible during its advancement.)
Complications | baseline
  A complication is defined as participants puncturing the arterial vessel of the simulator
Success of the procedure | 10 minutes from the baseline
  Procedure will be considered successful if participants will be able to insert the guidewire in a 10 minutes timeframe

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Veneto, Italy